CLINICAL TRIAL: NCT00623805
Title: A Randomized, Multicenter Phase III Trial to Assess the Efficacy and Safety of Bevacizumab and Capecitabine as Maintenance Treatment, After Initial Combination Treatment With Capecitabine, Oxaliplatin and Bevacizumab in Patients With Metastatic Colorectal Adenocarcinoma
Brief Title: A Study of Avastin (Bevacizumab) and Xeloda (Capecitabine) as Maintenance Treatment in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21440
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin

ARMS (2):
- Bevacizumab+capecitabine+oxaliplatin (Active Comparator): Participants received bevacizumab 7.5 mg/kg intravenously (IV) on Day 1 of each 3-week cycle + oxaliplatin 130 mg/m^2 IV on Day 1 of each 3-week cycle + capecitabine 1000 mg/m^2 orally twice a day on Days 1-14 of each 3-week cycle until disease progression.
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Oxaliplatin
- Bevacizumab(B)+capecitabine(C)+oxaliplatin followed by B+C (Experimental): Participants received bevacizumab 7.5 mg/kg intravenously (IV) on Day 1 of each 3-week cycle + oxaliplatin 130 mg/m^2 IV on Day 1 of each 3-week cycle + capecitabine 1000 mg/m^2 orally twice a day on Days 1-14 of each 3-week cycle for 6 cycles followed by bevacizumab 7.5 mg/kg intravenously (IV) on Day 1 of each 3-week cycle + capecitabine 1000 mg/m^2 orally twice a day on Days 1-14 of each 3-week cycle until disease progression.
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was supplied as a solution in single-use vials.
  Other Names: Avastin
Drug: Capecitabine — Capecitabine was supplied as film-coated tablets.
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin was supplied as a lyophilized powder in vials.
  Other Names: Eloxatin

SUMMARY:
This 2 arm study assessed the efficacy and safety of maintenance treatment with Avastin (bevacizumab) + Xeloda (capecitabine), after initial treatment with Xeloda + oxaliplatin + Avastin, in patients with metastatic colorectal cancer. Patients were randomized into one of 2 groups to receive 1) Xeloda + oxaliplatin + Avastin until disease progression or 2) Xeloda + oxaliplatin + Avastin for 6 3-week cycles, followed by Xeloda + Avastin until disease progression. Xeloda was administered at a dose of 1000 mg/m^2 orally twice a day on days 1-14 of each cycle, oxaliplatin at a dose of 130 mg/m^2 intravenously (iv) on day 1 of each cycle, and Avastin at a dose of 7.5 mg/kg iv on day 1 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age.
* Histologically confirmed colon or rectal cancer, with unresectable metastatic disease.
* At least 1 measurable lesion.
* Outpatient, with Eastern Cooperative Oncology Group (ECOG) Performance Status = 0-1.

Exclusion Criteria:

* Previous treatment with Avastin.
* Previous systemic treatment for advanced or metastatic disease.
* clinically significant cardiovascular disease.
* Daily chronic treatment with high doses of aspirin (> 325 mg/day) or non-steroidal anti-inflammatory drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Turkey (Türkiye) (5):
  - Ankara
  - Gaziantep
  - Istanbul
  - Izmir
  - S?hhiye, Ankara

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab+Capecitabine+Oxaliplatin | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C
Started | 62 | 61
Completed | 42 | 39
Not Completed | 20 | 22
Not completed — Adverse Event | 9 | 6
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 3 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Reason not Specified | 3 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants with a least 1 post-randomization efficacy assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab+Capecitabine+Oxaliplatin | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (11.2) | 57.6 (11.3) | 57.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 39 | 38 | 77

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the first administration of study drug to the first documented disease progression or death, whichever occurs first. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the unequivocal progression of existing non-target lesions. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions at Baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter for all target lesions will be calculated and reported as the Baseline sum longest diameter.
Time Frame: Baseline to the end of the study (up to 4 years, 2 months)
Population: Intent-to-treat population: All randomized participants who had at least 1 post-randomization efficacy assessment.
Measure: Mean (Standard Error); unit: Months
Arm/Group | Bevacizumab+Capecitabine+Oxaliplatin | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C
Number analyzed (Participants) | 62 | 61
Months | 9.0 (0.7) | 12.6 (1.0)

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the first administration of study drug to death.
Time Frame: Baseline to the end of the study (up to 4 years, 2 months)
Population: Intent-to-treat population: All randomized participants who had at least 1 post-randomization efficacy assessment.
Measure: Mean (Standard Error); unit: Months
Arm/Group | Bevacizumab+Capecitabine+Oxaliplatin | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C
Number analyzed (Participants) | 62 | 61
Months | 21.0 (1.3) | 25.4 (1.7)

3. Secondary Outcome: Percentage of Participants With a Complete Response or a Partial Response
Description: A complete response was defined as the disappearance of all target lesions. A partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the Baseline sum longest diameter. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions at Baseline. All other lesions (or sites of disease) should be identified as non-target lesions. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter for all target lesions will be calculated and reported as the Baseline sum longest diameter.
Time Frame: Baseline to the end of the study (up to 4 years, 2 months)
Population: Intent-to-treat population: All randomized participants who had at least 1 post-randomization efficacy assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab+Capecitabine+Oxaliplatin | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C
Number analyzed (Participants) | 62 | 61
Percentage of participants | 53.2 | 59.0

4. Secondary Outcome: Time Until a Complete Response or a Partial Response
Description: Time until a complete response or a partial response was defined as the time from the first administration of study drug until the first complete response or partial response.
Time Frame: Baseline to Month 13
Population: Intent-to-treat population: All randomized participants who had at least 1 post-randomization efficacy assessment. Only participants with a complete response or a partial response were included in the analysis.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Bevacizumab+Capecitabine+Oxaliplatin | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C
Number analyzed (Participants) | 33 | 36
Months | 3.5 (2.8) | 2.9 (2.0)

5. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the first complete response or partial response until disease progression or death. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the unequivocal progression of existing non-target lesions. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions at Baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter for all target lesions will be calculated and reported as the Baseline sum longest diameter.
Time Frame: Baseline to the end of the study (up to 4 years, 2 months)
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Participants With Metastatic Lesions Previously Considered Inoperable Who Became Operable and Underwent Surgery
Time Frame: Baseline to the end of the study (up to 4 years, 2 months)
Population: Intent-to-treat population: All randomized participants who had at least 1 post-randomization efficacy assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab+Capecitabine+Oxaliplatin | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C
Number analyzed (Participants) | 62 | 61
Percentage of participants | 58.1 | 54.1

7. Secondary Outcome: Percentage of Participants With a R0 Resection
Description: An R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.
Time Frame: Baseline to the end of the study (up to 4 years, 2 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safety population: All participants who received at least 1 dose of study drug.
Arm/Group | Bevacizumab+Capecitabine+Oxaliplatin | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C
Serious Adverse Events (participants affected / at risk) | 12/62 | 21/61
Other Adverse Events (participants affected / at risk) | 62/62 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Capecitabine+Oxaliplatin (N=62) | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C (N=61)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Acute renal failure (Renal and urinary disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Clinical worsening (General disorders) | 0 | 2
Decreased breath sounds on right lower zone (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Defence, distension and rigidity in abdomen (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 2
Difficulty in breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Febrile neutropenia (Infections and infestations) | 0 | 1
General situational failure (General disorders) | 0 | 1
Laryngeal edema (Immune system disorders) | 0 | 1
H1N1 infection (influenza) (Infections and infestations) | 1 | 0
High level of tiredness (General disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Neutropenic fever (Infections and infestations) | 1 | 0
Rapid advanced dyspnea and cyanosis (Cardiac disorders) | 0 | 1
Rectovaginal fistule (Gastrointestinal disorders) | 0 | 1
Severe backache, shivering (General disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Capecitabine+Oxaliplatin (N=62) | Bevacizumab(B)+Capecitabine(C)+Oxaliplatin Followed by B+C (N=61)
Nausea (Gastrointestinal disorders) | 27 | 17
Vomiting (Gastrointestinal disorders) | 24 | 16
Weakness (General disorders) | 24 | 18
Anorexia (Gastrointestinal disorders) | 17 | 13
Diarrhea (Gastrointestinal disorders) | 24 | 17
Neuropathy (Nervous system disorders) | 25 | 25
Hemifacial spasm (Vascular disorders) | 23 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.